CLINICAL TRIAL: NCT00754117
Title: Early Response Assessment in Patients With Diffuse Large B-cell Lymphoma Using 18-fluoro-2-deoxyglycose Positron Emission Tomography (FDG-PET)
Brief Title: Early Response Assessment in Diffuse Large B-Cell Lymphoma (DLCL) Patients by 18-fluoro-2-deoxyglycose Positron Emission Tomography (FDG-PET)
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0801009588
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: diffuse large b cell lymphoma; newly diagnosed
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: All patients

SUMMARY:
Newly diagnosed DLCL patients will have baselne FDG-PET as part of initial staging (PET-1). Patients will then undergo 2 cycles of chemotherapy with R/CHOP. 14 to 21 days following cycle 2 of R/CHOP, patients will undergo repeat FDG-PET scan (PET-2). They will then complete therapy as planned. Following completion of therapy, standard response assessment will be performed, including CT scans of the chest, abdomen and pelvis and FDG-PET scan (PET-3).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of CD20+ diffuse large B cell lymphoma (LBCL) of any stage, including subtypes mediastinal large B cell, centroblastic, immunoblastic, T cell rich B cell and anaplastic B cell lymphoma
* Patients must have received no prior anti-lymphoma therapy.
* Age >18 years.
* Patients must have a treatment plan to include R/CHOP or R/CHOP followed by radiotherapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have known HIV infection.
* Patients who are, in the opinion of their treating oncologist, unable to undergo R/CHOP chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed diffuse large b cell lymphoma patients planning to receive 6-8 cycles of R/CHOP chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2012-12-08 (Actual)

PRIMARY OUTCOMES:
evaluating the predictive value of a positive PET scan early in the course of standard chemotherapy | after 2 cycles of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Elstrom, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States